CLINICAL TRIAL: NCT01421524
Title: A Phase 1a/1b, Multi-center, Open-label, Dose Finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the Pleiotropic Pathway Modifier CC-122 Administered Orally to Subjects With Advanced Solid Tumors, Non-Hodgkin's Lymphoma, or Multiple Myeloma.
Brief Title: Study of CC-122 to Evaluate the Safety, Tolerability, and Effectiveness for Patients With Advanced Solid Tumors, Non-Hodgkin's Lymphoma, or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-ST-001; U1111-1203-5132 (Registry Identifier: WHO)
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Pleiotropic Pathway Modifier; Glioblastoma; Lymphoma; Primary Central Nervous System Lymphoma
Keywords: Neoplasm; Malignancy; Carcinoma; Lymphoma; Multiple Myeloma; DNA-PK inhibitor; Advanced Solid Tumors; Glioblastoma multiforme; Hepatocellular Carcinoma; Diffuse large B-cell lymphoma; Mantel Cell Lymphoma; Advanced unresectable Solid Tumors; Primary CNS Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Glioblastoma; Lymphoma; Neoplasms; Carcinoma; Carcinoma, Hepatocellular | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CC-122 MM-2 (Experimental): A new MM cohort (MM-2) will be enrolled in order to evaluate tolerability, safety and preliminary efficacy of the CC-122 formulated capsule given on an intermittent schedule (5/7 days per week) in 2 parallel dose escalation cohorts (MM-2a and MM-2b, respectively) (DEX) in Pomalidomide naïve subjects
  Interventions: Drug: CC-122
- CC-122- DLBCL-2 (Experimental): A new DLBCL cohort (DLBCL-2) in order to evaluate intermittent schedules of CC-122 (5 continuous days out of 7 days per week [5/7 days] and/or 21 continuous days out of 28 days per cycle [21/28 days]). Doses to be explored include 4 mg and 5 mg on an intermittent schedule using the 3+3 design described in Part A in order to establish an MTD for the intermittent dosing schedules. Following dose escalation, one or more intermittent dosing schedules may be expanded at or below the new intermittent schedule MTD in at least 20 total subjects per dosing schedule.
  Interventions: Drug: CC-122
- CC-122- GBM-2 (Experimental): A new GBM cohort (GBM-2) in order to evaluate doses of CC-122 above the 3 mg QD MTD determined in all comers in Part A. CC-122 dose will increase in 1 mg increments starting with 4 mg daily on a continuous schedule using the 3+3 design described in Part A in order to establish an MTD specific for GBM subjects. Following dose escalation, the cohort will be expanded at or below the new MTD in up to 20 total subjects.
  Interventions: Drug: CC-122
- Primary Central Nervous System Lymphoma (PCNSL) (Experimental): During dose expansion of selected intermittent schedules, an additional cohort of up to 10 subjects with PCNSL will also be explored at the same dose and schedule as DLBCL to confirm some safety and preliminary efficacy signal
  Interventions: Drug: CC-122

INTERVENTIONS:
Drug: CC-122 — CC-122 dose in both arms will increase by 1 mg increments starting with 3 mg 5/7 days using the 3+3 design in dose escalation phase. A dose-level -1, with a starting dose of 2mg, may also be evaluated if the opening dose level is not tolerated. At all dose levels in MM-2b arm, DEX will be combined with CC-122 at a starting dose dependent on the subject's age: for subjects who are ≤ 75 years of age, DEX 40 mg/day will be given on Days 1, 8, 15 and 22 of a 28-day cycle and for subjects who are > 75 years of age, DEX 20 mg/day will be given on Days 1, 8, 15 and 22 of a 28-day cycle. Approximately 33 subjects will be enrolled in the dose escalation phase (15 in each treatment arm). An additional intermittent schedule of 21/28 days may be evaluated per Safety Review Committee (SRC) decision. Following dose escalation, one or two arms will be expanded at or below the MTD in up to 28 subjects (14 subjects in each arm).
  Arms: CC-122 MM-2
Drug: CC-122 — One or more intermittent schedules of CC-122 either given 5 continuous days out of 7 per week (5/7 days) or 21 continuous days out of 28 days per cycle (21/28 days). Following dose escalation, one or more of these intermittent schedules will be evaluated at a starting dose of 4 mg.
  Arms: CC-122- DLBCL-2
Drug: CC-122 — Dose escalation on a continous schedule will be evaluated at a starting dose of 4 mg. Specifically, dose levels with 1 mg increments (eg 4mg, 5mg, 6mg etc.) will be evaluated using a 3+3 design as detailed in Part A of the protocol .
  Arms: CC-122- GBM-2
Drug: CC-122 — Up to 10 subjects with relapsed or refractory PCNSL will be enrolled to a PCNSL cohort to evaluate intermittent schedules of CC-122 and to further explore preliminary signals of efficacy and biomarker hypotheses.
  Arms: Primary Central Nervous System Lymphoma (PCNSL)

SUMMARY:
The main purpose of this first in human study with CC-122 is to assess the safety and action of a new class of experimental drug (Pleiotropic Pathway Modulator) in patients with advanced tumors unresponsive to standard therapies and to determine the appropriate dosing level and regimen for later-stage clinical trials.

DETAILED DESCRIPTION:
This trial is enrolling additional Multiple Myeloma (MM) subjects in a separate cohort defined as MM-2 to evaluate tolerability, safety and preliminary efficacy of CC-122 formulated capsule alone or in combination with DEX on intermittent dosing schedule (5 of 7 days of the week) in Pomalidomide-naïve subjects. Preliminary efficacy data in Multiple Myeloma subjects, warrants further exploration of CC-122 in MM on intermittent schedules to assess if dose intensity and tolerability can be improved. Initially, patients will be treated with oral CC-122 for one month. During this time, various tests (involving blood and urine collections, ECGs, etc) will be performed. Those whose tumors stabilize or regress may continue receiving treatment for as long as they benefit from CC-122. Different dose levels of CC-122 will be tested in a dose-rising study design.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
2. Men and women, 18 years or older, with histologically or cytologically-confirmed, advanced solid tumors, Non-Hodgkin Lymphona (NHL), Multiple Myloma (MM), or advanced unresectable solid tumors limited to the tumor types below.

   1. Subjects who have progressed on (or not been able to tolerate) standard anticancer therapy or for whom no standard anticancer therapy exists. Must have disease that is objectively measurable
   2. Measurable disease criteria:

      * Subjects with Glioblastoma multiforme (GBM) do not have to have objectively measurable disease at entry.
      * For MM, Diffuse large B-cell lymphoma (DLBCL): Subjects must have disease that is objectively measurable, measurable levels of myeloma paraprotein in serum (> 0.5 g/dL) or urine (> 0.2 g excreted in a 24-hour collection sample) for MM and measurable disease by Internatonal Working Group (IWG) for NHL (with at least one measurable lesion's longest diameter ≥ 2cm).
      * For Primary Central Nervous System (CNS) Lymphoma (PCNSL): Subjects must have disease that is objectively measurable by International Workshop to Standardize Baseline Evaluation and Response Criteria in Primary CNS Lymphoma, Cerebrospinal Fluid (CSF) cytology (in case of leptomeningeal only disease), or vitreal aspiration cytology and/or retinal photographs (in case of ocular lymphoma).
3. Tumor specific inclusion criteria:

   * DLBCL-2 cohort:

     * Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1.
     * Histologically proven diffuse large B-cell non-Hodgkin's lymphoma
     * Must have progressed following or have been unable to tolerate at least one prior anthracycline or alkylating agent containing regimen (with or without anti-CD20).
     * Platelets ≥ 60 x 109/L.
   * For PCNSL cohort:

     * ECOG Performance Status of ≤ 2
     * Recurrent/refractory CNS non-Hodgkin's lymphoma involving CNS (Brain, Cerebrospinal fluid (CSF) or intraocular compartments)
     * Stable dose of glucocorticoids pre-therapy. If patients are receiving glucocorticoids, the dose should not increase during the 96 hours prior to initiation of therapy.
     * ECOG Performance Status of ≤ 2.
   * For glioblastoma multiforme (GBM-2) cohort:

     * ECOG Performance Status of ≤ 2
     * Primary GBM or gliosarcoma
     * ECOG Performance Status of ≤ 2.
     * Has received prior treatment including radiation and chemotherapy, with radiation completed > 12 weeks prior to Day 1 (or ≥ 4 weeks if the recurrence is outside of the prior radiation field).
     * Progression of disease after last therapy demonstrated by RANO criteria
     * No prior therapy with Avastin
     * No prior or scheduled Gliadel® wafer implant unless area of assessment and planned resection is outside the region previously implanted.
     * No prior interstitial brachytherapy or stereotactic radiosurgery unless area of assessment and planned resection is outside the region previously treated.
     * No enzyme-inducing anti-epileptic drugs (EIAED) such as carbamazepine, phenytoin, phenobarbital, or primidone within 14 days before Day 1.
     * Able to undergo repeated magnetic resonance imaging (magnetic resonance imaging (MRI), computed tomography (CT) scans).
     * Availability of adequate Formalin-fixed, paraffin embedded (FFPE) archival tumor material.
     * Platelets (plt) ≥ 100 x 109/L.
   * For Multiple Myeloma cohort

     * ECOG Performance Status of ≤ 1.
     * Have a documented diagnosis of multiple myeloma and have relapsed and refractory disease.
   * Measurable levels of myeloma paraprotein (M-protein) in serum (> 0.5 g/dL) or urine (> 0.2 g excreted in a 24-hour collection sample).

     * Patients must have received at least 2 prior therapies.
     * Patients must have relapsed after having achieved at least stable disease for at least one cycle of treatment to at least one prior regimen and then developed PD.
     * Patients must also have documented evidence of PD during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry (refractory disease).
     * Patients must have also undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of a proteosome inhibitor (either in separate regimens or within the same regimen).
     * Must be Pomalidomide naïve.
   * Last dose of therapeutic glucocorticosteroids given greater than 14 days prior to start of study treatment.
   * Platelets (plt) ≥ 75 x 109/L in subjects in whom < 50% of bone marrow mononuclear cells are plasma cells or ≥ 30 x 109/L in subjects in whom ≥ 50% of bone marrow mononuclear cells are plasma cells.
4. At least 4 weeks from last dose of therapeutic glucocorticosteroids. Adrenal replacement doses of glucocorticosteroids (up to the equivalent of 10 mg daily prednisone) are allowed.
5. Biopsies (DLBLC, MM): Diagnostic archival FFPE (either in tumor blocks or sectioned/mounted specimens) may be submitted in lieu of a pre-study research biopsy if it has been obtained no more than 1 year prior to enrollment and only after discussion with the Celgene Medical Monitor
6. If not specified above as tumor specific parameter subjects must have the following laboratory and hematologic parameters as follows:

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if received pegfilgrastim).
   2. Hemoglobin (Hgb) ≥ 9 g/dL.
   3. Platelets (Plt) ≥100 x 109/L.
   4. Potassium within normal limits or correctable with supplements.
   5. AST/SGOT and ALT/SGPT ≤ 3 x upper limit of normal (ULN) or ≤ 5.0 x ULN if liver tumor is present.
   6. Serum creatinine ≤ ULN (with value applied to Cockcroft-Gault equation) or 24 hour clearance ≥ 50mL/min.
   7. Negative serum pregnancy test in females of childbearing potential

Exclusion Criteria:

1. History of other carcinomas within the last 5 years except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer with a current Prostate-specific antigen (PSA) of <1.0 mg/dL on 2 evaluations at least 3 months apart; the most recent evaluation must be no more than 4 weeks prior to Day 1 of the study drug, or other malignancies that were completely resected or treated Stage 1/2 lesions currently in complete remission.
2. Symptomatic central nervous system metastases (excluding Glioblastoma multiforrme (GBM) and Primary Central Nervous System Lymphoma (PCNSL). Subjects with brain metastases that have been previously treated and are stable for 6 weeks are allowed.
3. Known symptomatic acute or chronic pancreatitis.
4. Any peripheral neuropathy ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade 2.
5. Persistent diarrhea or malabsorption ≥ NCI CTCAE grade 2, despite medical management.
6. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiography (ECHO).
   2. Complete left bundle branch, or bifasicular block.
   3. Congenital long QT syndrome.
   4. Persistent or uncontrolled ventricular arrhythmias or atrial fibrillation.
   5. QTcF > 460 msec on screening Electrocardiography (ECG) (mean of triplicate recordings).
   6. Unstable angina pectoris or myocardial infarction ≤ 3 months prior to starting CC-122.
   7. Troponin-T value > 0.4 ng/ml or BNP >300 pg/mL.

      ° Subjects with baseline troponin-T >Upper Limit of Normal (ULN) or B-type Natriuretic Peptide (BNP) >100 pg/mL are eligible but must have cardiologist evaluation prior to enrollment in the trial for baseline assessment and optimization of cardioprotective therapy.
   8. Other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension (blood pressure ≥ 160/95 mmHg).
7. Other concurrent severe and/or uncontrolled concomitant medical conditions (eg, active or uncontrolled infection or renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol.
8. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy.
9. Major surgery ≤ 2 weeks prior to starting study drug or still recovering from post operative side effects.
10. Women who are pregnant or breast feeding. Adults of reproductive potential not employing two forms of birth control as per Pregnancy Prevention Risk Management Plan.
11. Known Human immunodeficiency virus (HIV) infection.
12. Known chronic hepatitis B or C virus (HBV/HCV) infection, unless comorbidity in subjects with Hepatocellular carcinoma (HCC).
13. Status post solid organ transplant.
14. Less than 100 days for subjects receiving autologous hematologic stem cell transplant (HSCT); or 6 months for subjects receiving allogenic HSCT or either transplant type, if otherwise not fully recovered from HSCT related toxicity.
15. For MM-2 cohort only: Hypersensitivity (eg, Rash Grade 3 or 4) to thalidomide, lenalidomide, or dexamethasone (MM-2b).
16. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
17. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
18. Any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to approximately Day 28
  Dose-limiting toxicities (DLTs) will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE):
  * A clinically relevant AE that is suspected to be related to CC-122 and starts ≤ 30 days of first dose (Cycle 1) and ≥ grade (Gr) 3 except for Alopecia, Gr3 rash of the acneiform or maculopapular type < 4 daysduration , Gr 3 diarrhea or vomiting lasting< 72 hours
  * Clinically relevant laboratory abnormality suspected to be related to CC-122 and that commences within 30 days of first dose and ≥ Gr3.
  * Hematological toxicities as follows: Any febrile neutropenia (NP), Gr4 NP > 7 days, Gr 4 thrombocytopenia > 24 hours, Any Gr 3/4 thrombocytopenia with clinically significant bleeding.
  * Gr 4 liver function tests (LFTs) or Gr 3 ALT with ≥ Gr2 bilirubin
  * Any AE suspected to be CC-122 related and necessitating dose reduction during Cycle 1.
Pharmacokinetics- Cmax | Up to day 22
  Maximum observed concentration in plasma (Cmax)
Pharmacokinetics- AUC | Up to day 22
  Area under the concentration-time curve
Pharmacokinetics- tmax | Up to day 22
  Time to maximum concentration
Pharmacokinetics- t1/2 | Up to day 22
  Terminal half-life
Pharmacokinetics- CL/F | Up to day 22
  Apparent total body clearance
Pharmacokinetics- Vz/F | Up to day 22
  Apparent volume of distribution
Non-tolerated dose (NTD) | Up to day 28
  Is defined as the dose level at which ≥2 out of 6 evaluable subjects in any dose cohort with DLT.
Maximum Tolerated Dose (MTD) | Up to day 28
  Is defined as the last dose level below the NTD with ≤1 out of 6 evaluable subjects with DLT) during Cycle (C) 1.

SECONDARY OUTCOMES:
Response Rate | up to approximately 6 months
  The response rate of each tumor types based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1), International Workshop Criteria (IWC) for Non-Hodgkin's Lymphoma (NHL), International Uniform Response Criteria for Multiple Myeloma (IURC), or Responses Assessment for Neuro-Oncology (RANO) working group for Glioblastama multiforme (GBM)
Tissue concentration of CC-122 | up to approximately 6 months
  Tissue concentration of CC-122 in salvage resection specimens from subjects with GBM (CNS primary tumor) or in cerebrospinal fluid (CSF) from subjects undergoing lumbar puncture.
6-month progression free survival (PFS) rate for GBM chort | Up to approximately 6 months
  The primary efficacy variable for GBM chohort is 6-month progression free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (17):
  - City of Hope Cancer Center, Duarte, California
  - UCLA Neuro-Oncology Program, Los Angeles, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey University, New Brunswick, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Local Institution - 020, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - MUSC Rheumatology and Immunology Dept., Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Sarah Cannon Research Institute Drug Development Unit, Nashville, Tennessee
  - Texas Oncology, PA - Dallas 75246, Dallas, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Swedish Medical Center Cancer Institute Research, Seattle, Washington
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington
- Belgium (2):
  - Local Institution - 401, Brussels
  - Local Institution - 400, Leuven
- France (5):
  - Local Institution - 202, Caen
  - Local Institution - 201, Marseille Le Cedex
  - Local Institution - 205, Pierre-Bénite
  - Local Institution - 203, Toulouse
  - Local Institution - 200, Villejuif
- Italy (6):
  - Local Institution - 303, Bologna
  - Local Institution - 305, Bologna
  - Local Institution - 300, Milan
  - Local Institution - 302, Napoli, Campania
  - Local Institution - 304, Roma
  - Local Institution - 301, Rozzano (MI)
- Spain (9):
  - Local Institution - 103, Badalona (Barcelona)
  - Local Institution - 105, Barcelona
  - Local Institution - 101, Barcelona
  - Local Institution - 104, Madrid
  - Local Institution - 102, Madrid
  - Local Institution - 106, Pamplona
  - Local Institution - 108, Salamanca
  - Local Institution - 107, Seville
  - Local Institution - 100, Valencia

REFERENCES:
- [Background] Rasco DW, Papadopoulos KP, Pourdehnad M, Gandhi AK, Hagner PR, Li Y, Wei X, Chopra R, Hege K, DiMartino J, Shih K. A First-in-Human Study of Novel Cereblon Modulator Avadomide (CC-122) in Advanced Malignancies. Clin Cancer Res. 2019 Jan 1;25(1):90-98. doi: 10.1158/1078-0432.CCR-18-1203. Epub 2018 Sep 10. PMID 30201761
- [Background] Cubillos-Zapata C, Cordoba R, Avendano-Ortiz J, Arribas-Jimenez C, Hernandez-Jimenez E, Toledano V, Villaescusa T, Moreno V, Lopez-Collazo E. CC-122 immunomodulatory effects in refractory patients with diffuse large B-cell lymphoma. Oncoimmunology. 2016 Sep 16;5(12):e1231290. doi: 10.1080/2162402X.2016.1231290. eCollection 2016. PMID 28255524
- [Background] Hagner P, et al. CC-122 Has Potent Anti-Lymphoma Activity through Destruction of the Aiolos and Ikaros Transcription Factors and Induction of Interferon Response Pathways. Presented at American Society of Hematology 2014, December 6-9, 2014, San Francisco, CA. Abstract No. 3035.
- [Derived] Carpio C, Bouabdallah R, Ysebaert L, Sancho JM, Salles G, Cordoba R, Pinto A, Gharibo M, Rasco D, Panizo C, Lopez-Martin JA, Santoro A, Salar A, Damian S, Martin A, Verhoef G, Van den Neste E, Wang M, Couto S, Carrancio S, Weng A, Wang X, Schmitz F, Wei X, Hege K, Trotter MWB, Risueno A, Buchholz TJ, Hagner PR, Gandhi AK, Pourdehnad M, Ribrag V. Avadomide monotherapy in relapsed/refractory DLBCL: safety, efficacy, and a predictive gene classifier. Blood. 2020 Mar 26;135(13):996-1007. doi: 10.1182/blood.2019002395. PMID 31977002
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com